CLINICAL TRIAL: NCT00861107
Title: Phase I/II Study of a Therapeutic Cancer Vacccine Created In-situ in Patients With Refractory or Metastatic Cancer
Brief Title: In-Situ Therapeutic Cancer Vaccine for Metastatic Cancer Combining AlloStim With Tumor Cryoablation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Dr. Michael Har-Noy, Immunovative Therapies, Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-002-CRYO
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Cancer
Keywords: Colorectal cancer; Breast Cancer; Melanoma; GI cancer; Prostate cancer; Kidney cancer; Lung cancer; all types metastatic cancer where at least one tumor lesion is accessable for percutaneous cryoablation
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Breast Neoplasms; Melanoma; Gastrointestinal Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: AlloStim-7 — intradermal injection once a week for 3 weeks
  Other Names: Priming Phase
Procedure: percutaneous tumor cryoablation — ablation of a tumor by percutaneous cryoablation under CT guidance
Biological: AlloStim-7 — intratumoral injection into cryoablated tumor lesion 1 hour after ablation
  Other Names: In-Situ Vaccine Phase
Biological: AlloStim8 or AlloStim-9 — intravenous infusion of AlloStim one week following ablation procedure. First cohort to receive 10^8 cell dose and if no toxicity dose escalates to 10^9 cell dose.
  Other Names: Immune activation phase

SUMMARY:
This is a Phase I/II study to investigate the feasibility of creating a personalized therapeutic cancer vaccine within the body. A vaccine contains a source of tumor antigen and an adjuvant. In this study, tumor antigen is generated by freezing a tumor by a minimally invasive percutaneous (through the skin) cryoablation procedure. The study drug, AlloStim, is injected into the ablated tumor to promote development of an anti-tumor immune response.

DETAILED DESCRIPTION:
This is a Phase I/II clinical study to investigate the feasibility of creating a personalized anti-tumor vaccine within the body of patients with advanced cancers. The aim of the study is to evaluate the safety of administration and anti-tumor effect of a vaccine protocol that has three separate phases. Cancer patients generally present with an immune response to cancer biased to a Th2 response, while a Th1 response is considered necessary for mediating anti-tumor immunity. The first step of the study consists of three (3) weekly intradermal priming doses of AlloStim. The aim of this step is to create Th1 immunity to the alloantigens in AlloStim, thus increasing the number of Th1 cells in circulation. The second step of the protocol involves the cryoablation of a selected tumor lesion followed by an intratumoral AlloStimTM injection. The aim of this step is to generate tumor-specific CTL killer cells in the circulation. The final step is an intravenous infusion of AlloStim. The aim of this step is to activate circulating Th1 cells, killer cells, and natural killer cells The further aim of this step is to create an inflammatory environment that can break-down the ability of the tumor to avoid an anti-tumor immune response.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Metastatic cancer refractory to at least one course of active chemotherapy or prior radiation therapy, including metastatic breast cancer, colorectal cancer, non-small cell lung cancer, ovarian or other gynecological cancer, prostate cancer, pancreatic or other GI cancer, melanoma, head or neck cancer or lymphoma/plasmacytoma.
* Measurable disease determined upon review of abdominal and/or chest CT scan within 60 days of evaluation for study inclusion with a target tumor lesion for cryoablation located in liver, kidney, bone, pancreas, lymph node, skin, neck or prostate deemed to be accessible for percutaneous access.
* Acceptable cryoablation procedure technique risk: the target tumor for ablation must have adequate distance from adjacent vasculature and other organs to permit safe application of cryoprobe (generally, more than a 2.5cm clearance of the cryoprobe from any vital structure such as the bowel, inferior vena cava, or aorta). The safety assessment of the cryoprobe placement will be made an attending radiologist based on imaging studies.
* Life expectancy >180 days
* No bevacizumab (Avastin®) within 6 weeks of planned cryoablation procedure
* ECOG status 0-1
* No concurrent medication known to interfere with platelet function or coagulation (e.g., aspirin, ibuprofen, clopidogrel, or warfarin) unless such medications can be discontinued for an appropriate time period based on the drug half-life and known activity (e.g., aspirin for 7 days) prior to cryoablation procedure
* No low molecular weight heparin preparations unless can be discontinued 8 hours prior to cryoablation
* At least 2 weeks since prior cytotoxic chemotherapy
* Absolute granulocyte count ≥ 1,200/mm3
* Platelet count ≥ 100,000/mm3
* PT/INR ≤ 1.5

  * INR correctable to ≤ 1.5 or a PT/PTT correctable to normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be monitored weekly prior to the cryoablation day 21 to assure INR is stable. However, heparin or warfarin must be withheld prior to cryoablation such that the above criteria are met.
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 mg/dL
* Total bilirubin ≤ 1.5 times normal
* Alkaline phosphatase ≤ 2.5 times normal (≤ 5 times normal if liver involvement)
* Aspartate aminotransferase (AST) or (SGOT) ≤ 2.5 times ULN
* Alanine aminotransferase (ALT) or (SGPT) ≤ 2.5 times ULN
* Not pregnant or lactating
* Patients with child bearing potential must agree to use adequate contraception
* No psychiatric or addictive disorders or other condition that, in the opinion of the investigator, would preclude study participation
* Study specific informed consent

Exclusion Criteria:

* Taking anticoagulant medication for concomitant medical condition (unless can be safely discontinued for cryoablation procedure)
* Prior allogeneic bone marrow/stem cell or solid organ transplant
* Chronic use (> 2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to > 10 mg/day of prednisone) within 30 days of the first day of study drug treatment

  * Topical and inhaled corticosteroids are permitted
* Concomitant autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, autoimmune thyroid disease, uveitis)
* Prior experimental cancer vaccine treatment (e.g., dendritic cell therapy, heat shock vaccine)
* Immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 3 months of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
evaluation of any drug-related toxicity associated with AlloStim administration as well as the reversibility of such toxicity. | 90 days

SECONDARY OUTCOMES:
evaluation of the anti-tumor effect of AlloStim administration | 90 days
evaluation of the immunological response to AlloStim administration | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Har-Noy, Study Director — Mirror Biologics, Inc.; Michael Berger, MD, Principal Investigator — Immunotherapy Clinical Associates, PC
Locations (1):
- Immunovative Clinical Research, Inc, Carlsbad, California, United States

REFERENCES:
- [Background] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631